CLINICAL TRIAL: NCT06192524
Title: OPTImal PHARMacological Therapy for Patients With Heart Failure: The OPTIPHARM-HF Registry
Acronym: OPTIPHARM-HF
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Azienda Socio Sanitaria Territoriale degli Spedali Civili di Brescia (Other)
Collaborators: Fondazione C.N.R./Regione Toscana "G. Monasterio", Pisa, Italy (Other Government); Centro Cardiologico Monzino (Other); A.O. Ospedale Papa Giovanni XXIII (Other); IRCCS Ospedale San Raffaele (Other); Azienda Ospedaliera Universitaria Senese (Other); Humanitas Research Hospital IRCCS, Rozzano-Milan (Other); Ospedale Policlinico San Martino (Other); Fondazione IRCCS Ca' Granda, Ospedale Maggiore Policlinico (Other); Fondazione IRCCS Policlinico San Matteo di Pavia (Other); Ospedali Riuniti di Foggia (Other); A.O.U. Città della Salute e della Scienza (Other); ASU Giuliano Isontina, Trieste (Unknown); Azienda Ospedaliera S. Maria della Misericordia (Other); IRCCS Policlinico S. Donato (Other); ASST Santi Paolo e Carlo (Other)
Responsible Party: Principal Investigator, Marco METRA, Marco Metra, Azienda Socio Sanitaria Territoriale degli Spedali Civili di Brescia
Other Study IDs: NP5441
Record Dates: First submitted 2023-12-21; First posted 2024-01-05 (Actual); Last update posted 2024-01-05 (Actual); Status verified 2023-12

CONDITIONS: Heart Failure
Keywords: GDMT; HFrEF; HFpEF; Clinical Outcomes
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years

SUMMARY:
Prospective, observational, multicenter, national study of adult patients with HF to assess prescription and adherence to evidence-based Guideline-Directed Medical Therapy (GDMT) in patients with Heart Failure (HF).

DETAILED DESCRIPTION:
Prospective, observational, multicenter, national study designed to evaluate the care and outcomes of patients with HF, to understand reasons for lack of implementation of evidence-based treatment and the impact of adherence to treatment on clinical outcomes in patients with HF across the full spectrum of left ventricular ejection fraction (LVEF).

The study will enroll consecutive patients with symptomatic HF, aged ≥ 18 years from at least 30 Italian tertiary HF care centers. Both outpatients and in-patients with chronic and acute decompensated HF will be consecutively recruited. Patients will be followed for a maximum duration of 24 months.

ELIGIBILITY:
Inclusion Criteria:

* Patients ≥ 18 years old
* Signed patient informed consent form (ICF)
* Diagnosis of chronic or acute decompensated HF according to ESC guidelines and the universal definition of HF.
* Receiving at least one drug for management of HF at study enrollment (including diuretics, β-blockers, angiotensin-converting enzyme inhibitors, angiotensin receptor blockers, aldosterone antagonists).

Exclusion Criteria:

* Planned participation or participation in a clinical trial;
* Life expectancy < 1 year because of non-cardiac causes;
* Previous heart transplant or left ventricular assist device implantation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Consecutive patients with symptomatic HF. Both outpatients and in-patients with chronic and acute decompensated HF will be consecutively recruited.
Sampling Method: Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2022-07-18 (Actual); Primary Completion 2024-10-01 (Estimated); Study Completion 2025-10-01 (Estimated)

PRIMARY OUTCOMES:
To describe the prevalence of use of GDMT, both as drugs administered and their dosing, defined according to target guidelines recommended doses, across the full spectrum of EF. | 1 year
  GDMT Prevalence and dosing

SECONDARY OUTCOMES:
To evaluate sequence of introduction of recommended GDMT, medications' up titration, when needed, maintenance of evidence-based treatment during follow-up | 1 year
  GDMT sequencing and up-titration
To describe GDMT implementation, dosing, and sequencing in specific HF population including de novo HF, worsening HF, advanced HF and HF with improved EF | 1 year
  GDMT in specific HF population
To assess cumulative rate of CV events and the impact on prognosis of GDMT and its doses. | 2 years
  * All-cause death
  * Cardiovascular death
  * Unplanned hospitalization for HF (including recurrent events)
  * Unplanned outpatient facility visits for HF where patient is treated with IV therapy
  * Heart transplantation or Ventricular Assist Device implantation
  * Non-fatal Myocardial Infarction (MI)
  * Non-fatal stroke
  * Atrial fibrillation events
  * ICD shock or hospitalization for ventricular arrhythmia
  * Hospitalization for acute kidney injury or other kidney disease event including dialysis or end-stage renal disease defined as eGFR < 15 mL/min/1.73 m2 or the need for renal replacement therapy.

CONTACTS AND LOCATIONS:
Overall Officials: Marco Metra, MD, Principal Investigator — ASST Spedali Civili; Riccardo M. Inciardi, MD, PhD, Principal Investigator — ASST Spedali Civili
Locations (1):
- ASST Spedali Civili, Brescia, Italy

IPD SHARING:
Plan to Share IPD: No